CLINICAL TRIAL: NCT03908372
Title: A Randomized Multicenter Phase II/III Study of Optimized Treatment Strategies for Stage II and III Nasopharyngeal Carcinoma
Brief Title: Optimized Treatment Strategies for Early and Medium Stage Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jun-Lin Yi, MD, professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC1950
Record Dates: First submitted 2019-03-31; First posted 2019-04-09 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Stage II, III; Nasopharyngeal Squamous Cell Carcinoma; Induction Chemotheray; Concurrent Chemoradiotherapy; Reduce Treatment Intensity
MeSH Terms: interventions — Docetaxel; Cisplatin; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Induction chemotherapy(IC)+IMRT (Experimental): Induction chemotherapy for two cycles, the patients with complete response will receive 60 Gy to the gross target volume of nasopharynx, partial response 64 Gy, and the absence of response will receive concurrent chemoradiotherapy as the same as CCRT arm
  Interventions: Drug: Docetaxel; Drug: Cisplatin; Radiation: IMRT
- Concurrent chemoradiotherapy(CCRT) (Active Comparator): cisplatin 100mg/m2 IV on d1 of each 21 days for two cycles at least and 70 Gy radiotherapy
  Interventions: Drug: Cisplatin; Radiation: IMRT

INTERVENTIONS:
Drug: Docetaxel — Induction CT: Docetaxel 75mg/m2 IV on d1, every 21 days for two cycles
  Other Names: Taxotere
  Arms: Induction chemotherapy(IC)+IMRT
Drug: Cisplatin — Induction chemotherapy:cisplatin 75mg/m2 IV on d1,every 21 days for two cycles.Concurrent chemoradiotherapy:cisplatin 100mg/m2 IV on d1 of each 21 days for at least two cycles during 70 Gy radiotherapy
  Other Names: DDP
Radiation: IMRT — IC+IMRT arm:the patients with complete response will receive 60Gy to the gross target volume of nasopharynx, partial response 64Gy, and the absence of response or stable will receive 70Gy. CCRT arm: 70Gy to the gross target volume of nasopharynx.
  Other Names: intensity-modulated radiotherapy

SUMMARY:
The purpose of this study is to optimize treatment strategies for patients with stage II and III nasopharyngeal carcinoma, reduce the side effects related to treatment and improve the quality of life.

DETAILED DESCRIPTION:
The data came from conventional studies showed that the distant metastases and toxicities associated with concurrent chemoradiotherapy were main problems for patients with clinical stage II and III nasopharyngeal carcinoma. However, inductive chemotherapy can decrease the likelihood of emergence of distant metastasis and reduce treatment related toxicities as previous studies showed.

The role of inductive chemotherapy in screening low-risk nasopharyngeal carcinoma for less treatment intensity is under-evaluated in the era of intensity-modulated radiotherapy (IMRT). we hope to find the optimized treatment strategies by reducing the intensity of treatment according to the treatment response of inductive chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Pathology confirmed nasopharyngeal squamous cell carcinoma.
* Aged 18 to 70 years old;
* Stage II-III (T1N1M0，T2-3N0-1M0) diseases according to 8th AJCC Staging and the shortest diameter of the largest lymph node involved is no more than 3cm;
* KPS≥70;
* Have measurable lesions on CT/MRI before treatment;
* Treatment for the first time;
* At least 6 months lifetime was expected;
* Adequate laboratory indexes, defined as follows: Hemoglobin > 120g/L, WBC > 4.0x10*9/L, Plt > 100x10*9/L < 2, all indexes of liver and kidney function ≤ 1.25 times of the institutional upper limit of normal value, no hearing loss;
* Can understand and sign the consent
* Have follow up condition

Exclusion Criteria:

* Past malignancies history (except for stage I non-melanoma skin cancer or cervical carcinoma in situ)
* Previously treatment for cancer
* Pregnant or breeding woman, female without contraception
* Enrolling in other drug trials
* Severe comorbidities including myocardial infarction, arrhythmia, cerebral vascular disease, ulceration disease, mental disease and uncontrolled diabetes
* Without follow up

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-06-15 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
progress free survival | 5 years

SECONDARY OUTCOMES:
overall survival | 5 years
local-regional control | 5 years
complete response | 13 weeks
  efficacy will be measured by RECIST1.1

CONTACTS AND LOCATIONS:
Overall Officials: Junlin Yi, professor, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Chinese Academy of Medical Sciences, Beijin, China

REFERENCES:
- [Background] Xu C, Sun R, Tang LL, Chen L, Li WF, Mao YP, Zhou GQ, Guo R, Lin AH, Sun Y, Ma J, Hu WH. Role of sequential chemoradiotherapy in stage II and low-risk stage III-IV nasopharyngeal carcinoma in the era of intensity-modulated radiotherapy: A propensity score-matched analysis. Oral Oncol. 2018 Mar;78:37-45. doi: 10.1016/j.oraloncology.2018.01.008. Epub 2018 Feb 20. PMID 29496056
- [Background] Liu YC, Wang WY, Twu CW, Jiang RS, Liang KL, Lin PJ, Lin JW, Lin JC. Comparison Long-term Outcome of Definitive Radiotherapy plus Different Chemotherapy Schedules in Patients with Advanced Nasopharyngeal Carcinoma. Sci Rep. 2018 Jan 11;8(1):470. doi: 10.1038/s41598-017-18713-z. PMID 29323141
- [Background] Yao JJ, Yu XL, Zhang F, Zhang WJ, Zhou GQ, Tang LL, Mao YP, Chen L, Ma J, Sun Y. Radiotherapy with neoadjuvant chemotherapy versus concurrent chemoradiotherapy for ascending-type nasopharyngeal carcinoma: a retrospective comparison of toxicity and prognosis. Chin J Cancer. 2017 Mar 6;36(1):26. doi: 10.1186/s40880-017-0195-6. PMID 28264724
- [Background] Xu C, Zhang LH, Chen YP, Liu X, Zhou GQ, Lin AH, Sun Y, Ma J. Chemoradiotherapy Versus Radiotherapy Alone in Stage II Nasopharyngeal Carcinoma: A Systemic Review and Meta-analysis of 2138 Patients. J Cancer. 2017 Jan 15;8(2):287-297. doi: 10.7150/jca.17317. eCollection 2017. PMID 28243333